CLINICAL TRIAL: NCT00347581
Title: A Randomized Clinical Trial of the Effectiveness of Base-in Prism Reading Glasses Vs. Placebo Reading Glasses for Symptomatic Convergence Insufficiency in Children
Brief Title: A Randomized Trial of Base-in Prism Reading Glasses Convergence Insufficiency in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pennsylvania College of Optometry (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: hms0304
Record Dates: First submitted 2006-07-03; First posted 2006-07-04 (Estimated); Last update posted 2006-07-04 (Estimated); Status verified 2005-01

CONDITIONS: Convergence Insufficiency
Keywords: convergence insufficiency; base-in prism; orthoptics; vision therapy
MeSH Terms: conditions — Ocular Motility Disorders

INTERVENTIONS:
Procedure: Base-in prism glasses for reading
Procedure: Placebo reading glasses

SUMMARY:
This study is designed to compare the use of special prism glasses to placebo treatment for children with symptomatic convergence insufficiency.

DETAILED DESCRIPTION:
The Base-in for Convergence Insufficiency Treatment Trial (BI-CITT) is a multi-center, placebo-controlled, masked, clinical trial designed to compare the benefits of base-in prism for patients with convergence insufficiency (CI).

The goals of this clinical trial are:

* To compare the effectiveness of Base-in prism and Placebo eyeglasses for the treatment of CI in children
* To study the long-term effect of these treatments for CI
* To identify factors that may be associated with successful treatment of CI with base-in prism

ELIGIBILITY:
Inclusion Criteria:

* Age: 9 to <19 years.
* Best corrected visual acuity of ≥20/25 in each eye at distance and near
* Willingness to wear eyeglasses or contact lenses to correct refractive error, if necessary
* Willingness to wear glasses for reading and other near work
* Exophoria at near at least 4 greater than at far
* Insufficient positive fusional convergence (fails Sheard's criterion)
* Receded near point of convergence of  6 cm break
* Random dot stereopsis appreciation using a 500 seconds of arc target.
* CI Symptom Survey score  16

Exclusion Criteria:

* Amblyopia (> 2 line difference in best corrected visual acuity between the two eyes).
* Constant strabismus
* History of strabismus surgery.
* Anisometropia  2D in any meridian between the eyes.
* Prior refractive surgery.
* Vertical heterophoria greater than 1 .
* Systemic diseases known to affect accommodation, vergence and ocular motility such as: multiple sclerosis, Graves thyroid disease, myasthenia gravis, diabetes, Parkinson disease.
* Any ocular or systemic medication known to affect accommodation or vergence (Anti-anxiety agents (Librium or Valium), Anti-arrhythmic agents (Cifenline or Cibenzoline), Anticholinergics (Motion sickness patch (scopolamine), Bladder spasmolytic drugs (Propiverine), Chloroquine, Phenothiazines (Compazine, Mellaril, or Thorazine), Tricyclic antidepressants (Elavil, Nortriptyline, or Tofranil)
* Accommodative amplitude <5 D in either eye as measured by the Donder's push-up method.
* Manifest or latent nystagmus.
* Developmental disability, mental retardation, attention deficit hyperactivity disorder (ADHD), or learning disability diagnosis in children that in the investigator's discretion would interfere with treatment.
* Household member or sibling already enrolled in the BI-CITT.
* Any eye care professional, ophthalmic technician, ophthalmology or optometry resident or optometry student.

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72
Dates: Start 2003-05; Study Completion 2004-08

PRIMARY OUTCOMES:
Symptom score on the Convergence Insufficiency Symptom Survey

SECONDARY OUTCOMES:
Near point of convergence
Positive fusional vergence at near

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Scheiman, OD, Study Chair — Pennsylvania College of Optometry
Locations (10):
- United States (10):
  - University of Alabama, Birmingham, College of Optometry, Birmingham, Alabama
  - Southern California College of Optometry, Fullerton, California
  - NOVA College of Optometry, Fort Lauderdale, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Indiana University College of Optometry, Bloomington, Indiana
  - State University of New York, College of Optometry, New York, New York
  - The Ohio State University, Optometry Coordinating Center, Columbus, Ohio
  - The Ohio State University, Columbus, Ohio
  - Eye Institute, Pennsylvania College of Optometry, Philadelphia, Pennsylvania
  - University of Houston, College of Optometry, Houston, Texas

REFERENCES:
- [Result] Scheiman M, Cotter S, Rouse M, Mitchell GL, Kulp M, Cooper J, Borsting E; Convergence Insufficiency Treatment Trial Study Group. Randomised clinical trial of the effectiveness of base-in prism reading glasses versus placebo reading glasses for symptomatic convergence insufficiency in children. Br J Ophthalmol. 2005 Oct;89(10):1318-23. doi: 10.1136/bjo.2005.068197. PMID 16170124
- [Derived] Scheiman M, Kulp MT, Cotter SA, Lawrenson JG, Wang L, Li T. Interventions for convergence insufficiency: a network meta-analysis. Cochrane Database Syst Rev. 2020 Dec 2;12(12):CD006768. doi: 10.1002/14651858.CD006768.pub3. PMID 33263359